CLINICAL TRIAL: NCT07230587
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Long-Term Efficacy of Butylphthalide in Patients With Minor Acute Ischemic Stroke (BLESS)
Brief Title: Butylphthalide for Long-term Efficacy in Minor Stroke Study
Acronym: BLESS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLESS; 2023ZD0504900 (Other Grant/Funding Number: National Science and Technology Major Project)
Record Dates: First submitted 2025-07-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Minor Stroke
Keywords: minor stroke; Butylphthalide
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide (Experimental): Butylphthalide 200 mg (oral soft capsules), three times daily for 12 months
  Interventions: Drug: Butylphthalide
- Placebo (Placebo Comparator): Placebo (matching oral soft capsules), three times daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Butylphthalide — Butylphthalide (NBP) is a neuroprotective agent derived from celery seed. It has demonstrated potential benefits in improving microcirculation, reducing oxidative stress, and protecting against neuronal injury in ischemic stroke. This study uses butylphthalide soft capsules (200 mg per dose) administered orally, three times daily for 12 months, to evaluate its long-term efficacy and safety in patients with minor acute ischemic stroke
  Other Names: 3-n-Butylphthalide; NBP
  Arms: Butylphthalide
Drug: Placebo — Matching placebo soft capsules, identical in appearance to butylphthalide capsules, administered orally at a dose of one capsule (200 mg equivalent) three times daily for 12 months. The placebo contains inactive ingredients without pharmacological effects and is used as a control to assess the efficacy and safety of butylphthalide in patients with minor acute ischemic stroke.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the long-term efficacy and safety of butylphthalide in patients with minor acute ischemic stroke (BLESS Trial).

A total of 1200 participants aged 40 to 80 years with a minor acute ischemic stroke confirmed by MRI will be enrolled. Participants will be randomly assigned in a 1:1 ratio to receive butylphthalide or placebo for 12 months.

The primary outcome is a hierarchical composite endpoint assessed at 12 months, including:

1. All-cause mortality
2. Stroke recurrence
3. Modified Rankin Scale (mRS) score ≥2
4. New MRI-confirmed infarcts
5. Change in Montreal Cognitive Assessment (MoCA) score from baseline

Secondary outcomes include additional functional, cognitive, and imaging-based assessments at 12 months.

This study aims to determine whether butylphthalide can improve long-term functional and cognitive outcomes in patients with minor ischemic stroke, contributing to better secondary stroke prevention strategies.

DETAILED DESCRIPTION:
1. Background and Rationale Minor acute ischemic stroke accounts for a significant proportion of all ischemic strokes and is associated with a substantial risk of recurrent stroke and cognitive impairment. Despite advances in secondary stroke prevention, effective long-term treatments targeting both functional recovery and neuroprotection remain limited. Butylphthalide, a compound originally derived from celery seed, has demonstrated neuroprotective, anti-inflammatory, and microcirculatory-enhancing effects in preclinical and clinical studies. Previous trials have suggested its potential benefits in improving neurological function and preventing stroke progression.

   The BLESS Trial (Butylphthalide for Long-term Efficacy in Minor Stroke Study) is designed to evaluate the long-term efficacy and safety of butylphthalide in patients with minor acute ischemic stroke, focusing on its impact on functional outcomes, cognitive performance, and neuroimaging markers.
2. Study Design and Methods

   This is a multicenter, randomized, double-blind, placebo-controlled trial that will enroll approximately 1200 participants across 50 sites in China. Participants will be randomized in a 1:1 ratio to receive: Butylphthalide soft capsules (200 mg, three times daily) for 12 months, or Matching placebo for 12 months.

   Participants will undergo regular follow-ups with comprehensive assessments of clinical, cognitive, and imaging parameters.
3. Primary Outcome Measure

A hierarchical composite endpoint assessed at 12 months using the Win Ratio method, prioritizing the following outcomes:

* All-cause mortality

  ②Stroke recurrence

  ③Modified Rankin Scale (mRS) score ≥2

  ④New MRI-confirmed infarcts

  ⑤Change in Montreal Cognitive Assessment (MoCA) score from baseline

  4.Secondary Outcome Measures
* All-cause mortality

  * Recurrent stroke

    * Modified Rankin Scale (mRS) score ≥2

      * MRI-confirmed new infarcts

        * Composite endpoint of ① + ② + ③

          * Composite endpoint of ① + ② + ③ + ④

            * Distribution of mRS scores ⑧ Change in MMSE score from baseline

              * Change in MoCA score from baseline

                * IADL score ⑪ Change in total Fazekas score of white matter hyperintensities from baseline ⑫ Change in white matter hyperintensity volume from baseline

                  ⑬ Change in DTI parameters from baseline

                  5. Statistical Analysis The Win Ratio method will be used for primary endpoint analysis, prioritizing mortality and severe disability outcomes. Secondary outcomes will be analyzed using Cox proportional hazards models, mixed-effects models, and logistic regression as appropriate. A significance level of P < 0.05 will be considered statistically significant.

                  6.Study Significance This study aims to determine whether butylphthalide can improve long-term functional and cognitive outcomes in minor stroke patients and provide a novel neuroprotective strategy for secondary stroke prevention. If successful, the findings could influence clinical guidelines for stroke management.

ELIGIBILITY:
1.Inclusion Criteria:

1. Age between 40 and 80 years old.
2. NIHSS score 0-5 at the time of stroke diagnosis, with MRI-confirmed acute ischemic infarct.
3. Time from stroke onset to enrollment ≤ 2 weeks.
4. Pre-stroke mRS score ≤ 1.
5. No prior diagnosis of cognitive impairment or dementia.
6. Informed consent must be voluntarily signed by the patient or their legal representative.

Exclusion Criteria:

1. Based on the TOAST classification, consider cardioembolic stroke, stroke of other determined etiology, or stroke of undetermined etiology.
2. Intracranial hemorrhagic diseases on imaging: hemorrhagic stroke, epidural hematoma, subarachnoid hemorrhage, etc. (If hemorrhagic transformation is present, eligibility is at investigator's discretion.)
3. Carotid artery stenosis > 50% requiring surgical intervention.
4. Systemic diseases causing cognitive impairment (e.g., endocrine diseases, vitamin deficiency, systemic autoimmune diseases).
5. Neurological disorders causing cognitive impairment, such as CNS infections, Creutzfeldt-Jakob disease, primary Parkinson's disease, traumatic brain injury, epilepsy, brain tumors.
6. Pre-stroke diagnosis of severe psychiatric disorders, including but not limited to depression, non-vascular cognitive impairment, or dementia (e.g., Alzheimer's disease, Parkinson's disease dementia, Lewy body dementia, frontotemporal dementia, drug or alcohol-induced cognitive impairment).
7. Severe hemiplegia and aphasia that significantly affect cognitive assessment.
8. Use of cognitive-enhancing drugs within 4 weeks before screening, including cholinesterase inhibitors (donepezil, rivastigmine, galantamine), NMDA receptor antagonists (memantine), sodium oligomannate (GV-971), or monoclonal antibodies (lecanemab, donanemab, aducanumab).
9. Severe liver disease (e.g., acute hepatitis, active chronic hepatitis, cirrhosis) or ALT/AST > 2× ULN.
10. Severe kidney disease or renal impairment (serum creatinine > 1.5× ULN).
11. Coagulation disorders or thrombocytopenia (platelet count < 100 × 10⁹/L).
12. Severe systemic diseases with an expected survival < 1 year.
13. Contraindications for MRI or inability to complete MRI scan.
14. Allergy to butylphthalide.
15. Pregnancy, lactation, or planned pregnancy.
16. Participation in another clinical trial within 30 days before randomization.
17. Deemed unsuitable for the study by the investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  The number of participants who experience all-cause mortality at 12 months. All-cause mortality includes death from any reason, such as cardiovascular, neurological, or other systemic causes.
Stroke recurrence | 12 months
  The number of participants who experience a recurrent stroke within 12 months. Recurrent stroke is defined as a new ischemic or hemorrhagic stroke, confirmed by neurological symptoms lasting ≥24 hours and neuroimaging evidence (MRI or CT)
Modified Rankin Scale (mRS) Score ≥2 | 12 months
  The proportion of participants with a modified Rankin Scale (mRS) score ≥2 at 12 months. The mRS is a widely used functional outcome measure that assesses the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with scores of 2 or higher indicating functional dependence.
New MRI-Confirmed Infarcts | 12 months
  The number of new infarcts confirmed by MRI at 12 months, compared to baseline. New infarcts are defined as newly developed ischemic lesions identified on diffusion-weighted imaging (DWI) or fluid-attenuated inversion recovery (FLAIR) sequences. A higher number of new infarcts indicates increased disease progression.
Change in Montreal Cognitive Assessment (MoCA) Score from Baseline | 12 months
  The change in Montreal Cognitive Assessment (MoCA) Score from baseline to 12 months. The MoCA is a cognitive screening tool that assesses multiple domains, including attention, concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
All cause mortality | 12 months
  The number of participants who experience all-cause mortality at 12 months. All-cause mortality includes death from any reason, such as cardiovascular, neurological, or other systemic causes.
Stroke Recurrence | 12 months
  The number of participants who experience a recurrent stroke within 12 months. Recurrent stroke is defined as a new ischemic or hemorrhagic stroke, confirmed by neurological symptoms lasting ≥24 hours and neuroimaging evidence (MRI or CT)
Distribution of Modified Rankin Scale (mRS) Scores | 12 months
  The distribution of mRS scores among participants at 12 months. The mRS assesses the degree of disability or dependence in daily activities following a stroke, ranging from 0 (no symptoms) to 6 (death). The distribution of scores across the treatment and control groups will be analyzed.
New MRI-Confirmed Infarcts | 12 months
  The number of new infarcts confirmed by MRI at 12 months, compared to baseline. New infarcts are defined as newly developed ischemic lesions identified on diffusion-weighted imaging (DWI) or fluid-attenuated inversion recovery (FLAIR) sequences.
Change in Mini-Mental State Examination (MMSE) Score from Baseline | 12 months
  The change in MMSE score from baseline to 12 months. The MMSE is a widely used cognitive screening tool that evaluates orientation, attention, memory, language, and visual-spatial skills. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Change in Montreal Cognitive Assessment (MoCA) Score from Baseline | 12 months
  The change in MoCA score from baseline to 12 months. The MoCA is a cognitive screening tool assessing attention, concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function
Change in Instrumental Activities of Daily Living (IADL) Score | 12 months
  The change in IADL score from baseline to 12 months. The IADL measures the ability to perform more complex daily activities required for independent living, including managing finances, medication adherence, cooking, and housekeeping. Higher scores indicate greater independence
Change in White Matter Hyperintensity (WMH) Fazekas Score from Baseline | 12 months
  The change in White Matter Hyperintensity (WMH) Fazekas Score from baseline to 12 months. The Fazekas scale is a validated measure of small vessel disease burden, ranging from 0 (no WMH) to 6 (severe WMH involvement)
Change in White Matter Hyperintensity Volume from Baseline | 12 months
  The change in WMH volume from baseline to 12 months, assessed using quantitative MRI analysis. This measure evaluates the impact of treatment on the progression of small vessel disease. A decrease in WMH volume suggests treatment efficacy.
Change in Diffusion Tensor Imaging (DTI) Parameters from Baseline | 12 months
  The change in DTI parameters from baseline to 12 months, including fractional anisotropy (FA) and mean diffusivity (MD). DTI is an MRI-based method for assessing white matter integrity and structural connectivity. Changes in FA and MD may reflect microstructural alterations associated with neuroprotection or disease progression.
Modified Rankin Scale (mRS) score ≥2 | 12 months
  The proportion of participants with a modified Rankin Scale (mRS) score ≥2 at 12 months. The mRS is a widely used functional outcome measure that assesses the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with scores of 2 or higher indicating functional dependence.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan Z, Zhao Y, Yang W, He S, Ding Y, Xu A. Efficacy and Safety of Adherence to dl-3-n-Butylphthalide Treatment in Patients With Non-disabling Minor Stroke and TIA-Analysis From a Nationwide, Multicenter Registry. Front Neurol. 2021 Sep 22;12:720664. doi: 10.3389/fneur.2021.720664. eCollection 2021. PMID 34630292
- [Result] Amarenco P, Lavallee PC, Monteiro Tavares L, Labreuche J, Albers GW, Abboud H, Anticoli S, Audebert H, Bornstein NM, Caplan LR, Correia M, Donnan GA, Ferro JM, Gongora-Rivera F, Heide W, Hennerici MG, Kelly PJ, Kral M, Lin HF, Molina C, Park JM, Purroy F, Rothwell PM, Segura T, Skoloudik D, Steg PG, Touboul PJ, Uchiyama S, Vicaut E, Wang Y, Wong LKS; TIAregistry.org Investigators. Five-Year Risk of Stroke after TIA or Minor Ischemic Stroke. N Engl J Med. 2018 Jun 7;378(23):2182-2190. doi: 10.1056/NEJMoa1802712. Epub 2018 May 16. PMID 29766771